CLINICAL TRIAL: NCT03203226
Title: The Feldenkrais Method for Improving Functioning and Body Balance in People With Intellectual Disability: a Randomized Clinical Trial
Brief Title: The Feldenkrais Method for People With Intellectual Disability
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of the Basque Country (UPV/EHU) (Other)
Responsible Party: Principal Investigator, JON TORRES UNDA, PRINCIPAL INVESTIGATOR, University of the Basque Country (UPV/EHU)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: M10/2015/151
Record Dates: First submitted 2017-06-27; First posted 2017-06-29 (Actual); Last update posted 2017-07-02 (Actual); Status verified 2017-06

CONDITIONS: Intellectual Disability
Keywords: Intellectual Disability; Feldenkrais Method; Short Physical Performance Battery; Stabilometry; Supported employment
MeSH Terms: conditions — Intellectual Disability

STUDY DESIGN:
Intervention Model Description: Participants will be recruited at a company which provides supported employment. The primary recruitment strategy will be the information provided to the potential participants and legal guardians by the medical staff of the company. Informed consent will be obtained from the participants and their legal guardians. Afterwards they will be randomly assigned (1:1 ratio) by centre through sealedopaque envelopes to either the control or the intervention group by coin-tossing sequence generation.
  It has been designed an experimental multicentre simple randomized study, with random allocation to a control group (CG) or to an experimental group (EG). This study is an open-label trial as the assessors who were experienced specialist in working with people with ID (psychologists, nurses, physicians, physiotherapists) are not blinded to group allocation.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- EXPERIMENTAL GROUP (Experimental): This protocol has an unique period or phase of 30 week. Experimental group will be composed by 30 volunteer who were previously randomly assigned to this group. This group will receive a intervention based on 30 1-hour session of Feldenkrais Method (1 hour per week).
  Interventions: Other: FELDENKRAIS METHOD (FM)
- CONTROL GROUP (No Intervention): This protocol has an unique period or phase of 30 week. Control group will be composed by 30 volunteer who were previously randomly assigned to this group. They will not receive any intervention.

INTERVENTIONS:
Other: FELDENKRAIS METHOD (FM) — They EG will receive the intervention of FM consisting of 30 lessons (1h-lesson per week; 30 weeks) verbal instructions provided by the therapist to participants. These instructions provide different options on how to perform a specific task with the purpose of leaving the decision on how to do the movement up to the performer, who has to focus on thinking, feeling, sensing and doing the movement as easily as possible.The lessons can be conducted sitting, standing or moving within a room.
  Arms: EXPERIMENTAL GROUP

SUMMARY:
Loss of functioning and age-related health problems tend to appear earlier in individuals with intellectual disability (ID) than in their non-disabled peers and due to this people with ID who are in employment tend to need to retire earlier, producing social, economic and health problems. The Feldenkrais method (FM) is a movement-based form of learning that enhances body balance and physical functioning. We hypothesized that the FM could be helpful to improve balance and functioning of employed people with ID.

DETAILED DESCRIPTION:
The aim of this study will be to determine the effects of a Feldenkraisn Method (FM) program in improving functionality and body balance in supported employed individuals with ID. To evaluate this effect, a total of subjects will participate in a longitudinal and clinical trial.

Sample size has been calculated to detect minimal significant effects on the variable of physical performance (SPPB): accepting an alpha risk of 0.05 and a beta risk of 0.20 in a bilateral contrast, 26 individuals are required in order to detect a difference equal to or greater than 1.5 unit in the SPPB (SD= 1.94). It has been increased the sample size in an additional 20% (losts during follow-up) and 5% (mortality). The resultant sample size is determinate in 32 individuals, who are equally randomized in both experimental and control groups.

Statistical analysis was performed using IBM SPSS Statistics for Windows (Version 22.0). Data were presented as mean ± standard deviation. Descriptive statistics were calculated for all outcome measures. Mean differences within the groups in the functional tests and stabilometric outcomes were estimated using paired sample t-tests, while mean differences between the groups in these variables were estimated using repeated measures analysis of variance. Differences were considered significant at p < 0.05. To determine the magnitude of the interactions between time and group, the effect size or µ2 was calculated as described by Cohen (1998) and interpreted as small (> 0.01 and < 0.06), moderate (≥ 0.06 and < 0.14) or large (≥ 0.14).

ELIGIBILITY:
Inclusion Criteria:

* Aged between 40 and 60 years old, with mild-moderate ID and able to follow FM classes in a group

Exclusion Criteria:

* Aged 40 or older than 60 years old, ID not classified as mild-moderate and absence of capacity for following FM classes in a group

Ages: 40 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2016-01-01 (Actual); Primary Completion 2016-12-28 (Actual); Study Completion 2017-01-30 (Actual)

PRIMARY OUTCOMES:
CHANGE FROM BASELINE PHYSICAL PERFORMANCE MEASURED BY SPPB (SCORE) AT 30 WEEKS | Participants are assessed at baseline (1 week before the intervention) and at 30 weeks.
  The Short Physical Performance Battery (SPPB) is a composite score of performance (0-12) based on 3 functional tasks. On each task, subjects can score between 0-4, with the higher values representing the best performance. Walking speed at a 4 m course is timed. Chair rise represented the time to complete 5 chair rises as quickly as possible. As a balance measure, standing balance score is used with responses ranging between 0-4. The sum of above mentioned three tasks provides the total SPPB score. Based on their subsequent risk for disability, mobility limitations have been characterized as being mild (score ≥10), moderate (score 7-9), and severe (score 4-6).

SECONDARY OUTCOMES:
Body height (cm) | Participants are assessed at baseline (1 week before the intervention) and at 30 weeks.
  Body height is measured (in cm) using a stadiometer (Marsden, T-226, UK) with the participant standing, wearing no shoes.
Body weight (kg) | Participants are assessed at baseline (1 week before the intervention) and at 30 weeks.
  Body weight is measured using a digital floor scale (Tanita, HD-314w, USA) with participants wearing light clothes and no shoes.
CHANGE FROM BASELINE STABILOMETRY (MM) (MM2) AT 30 WEEKS | Participants are assessed at baseline (1 week before the intervention) and at 30 weeks.
  Postural control is assessed with a static stabilometric platform (Winposture, Medicapteurs, FR) at an acquisition frequency of 50 Hz. Participants are asked to stand as still as possible with the eyes opened and bare foot during 60 sec. In order to ensure the same foot position for all the subjects, they are placed on the platform using a plastic device provided with this. Participants were instructed to look straight ahead at a mark placed onto the wall 2 m away at eye level. Data collection is initiated after participants adopted the required posture on the platform, stabilized their postural sway and signalled the experimenter that they are ready to begin. For security reasons, an assessor remains near the participant without touching or providing additional instructions during the test. Displacements of the centre of gravity are expressed in terms of sway area (mm2) and path length (mm).

CONTACTS AND LOCATIONS:
Overall Officials: JON TORRES, PHD, Principal Investigator — University of the Basque Country (UPV/EHU)

IPD SHARING:
Plan to Share IPD: No